CLINICAL TRIAL: NCT00367523
Title: Prevalence of Secondary Arterial Hypertension (PAH) in Patients With Sickle Cell Disease in Nigeria and the Role of HIV/AIDS and Endemic Parasitic Infections in the Natural History of Pulmonary Hypertension in Sickle Cell Disease
Brief Title: Pulmonary Hypertension in Patients With Sickle Cell Disease in Nigeria
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906189; 06-H-N189
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2017-09-28

CONDITIONS: Secondary Pulmonary Arterial Hypertension; Sickle Cell Disease; Pulmonary Hypertension
Keywords: Echocardiogram; Nigeria; Screening; Sickle Cell Disease; Genetics
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary

SUMMARY:
This study will explore how people with sickle cell disease (SCD) develop a complication called pulmonary hypertension (PHTN), a serious disease in which blood pressure in the lungs is higher than normal. PHTN is also caused by HIV, hepatitis C and schistosomiasis. Patients who have both SCD and one of these other infections may develop more severe PHTN. The number of Nigerians with SCD who also have PHTN is not known, nor is the cause of PHTN in this population. This study will examine genetic material in people with and without SCD to determine whether certain genes will allow doctors to predict which patients with SCD are likely to develop PHTN.

Nigerian males and females 10 years of age and older with or without SCD may be eligible for this study. Patients must have SS, SC, or SB thalassemia or other genotype; control subjects must have hemoglobin A or AS genotype.

Participants undergo a complete medical history and physical examination, blood tests, electrocardiogram (EKG), ultrasound tests of the heart and abdomen, and a 6-minute walk (distance test) to determine exercise capacity. Blood tests include screening for HIV, hepatitis B and C, schistosomiasis, hookworm and malaria. Patients who test positive for HIV, hepatitis B or C, schistosomiasis, hookworm or malaria are referred for treatment at Ahmadu Bello University Teaching Hospital in Zaria, Nigeria, and those who test negative for hepatitis B are referred for vaccination. Genetic tests focus on genes involved in SCD, PHTN, inflammation, blood vessel function and red blood cell function.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an autosomal recessive disorder and the most common genetic disease in the world. SCD is the most common inherited blood disorder in the United States, affecting 70,000 to 80,000 Americans. Secondary pulmonary arterial hypertension (PAH) has been shown to have a prevalence of 30% in patients with SCD with mortality rates of 40% at 40 months after diagnosis in the United States. The burden of disease of SCD is highest in Nigeria (West Africa) where approximately 4% of the 140 million people in that country are homozygous for SCD, but the prevalence and outcomes of pulmonary hypertension in Africa have not been investigated. Many known infectious risk factors for PAH are also highly prevalent in Nigeria, including Human Immuno Deficiency Virus/Acquired Immune Deficiency Syndrome (HIV/AIDS), malaria, chronic hepatitis B and C, schistosomiasis and hookworm. Our first clinical hypothesis is that interactions between these infectious complications and sickle cell related hemolysis would lead to an even higher prevalence of PAH in Nigeria. Our study is therefore designed to determine the prevalence of PAH in Nigerian patients with SCD using echocardiographic measurements of the tricuspid regurgitant jet velocity. We aim to determine the associations and epidemiological interactions that might lead to PAH, of endemic infectious disease co-morbidities, especially HIV/AIDS, with SCD by screening for these infectious diseases in control subjects and in SCD patients with and without PAH. Our second translational hypothesis is that genetic polymorphisms in candidate genes that regulate endothelial function and adhesion contribute to the development of PAH phenotype in African SCD patients. Using both candidate gene and genome wide association approaches, we will identify and selectively characterize single nucleotide polymorphisms (SNPs) in genes important for endothelial function, vascular inflammation and cardiac function (functional VCAM1 SNPs and steady state soluble VCAM-1 levels, SELP, SELE, SELL, ICAM1, ITGA4, and CD36, TGF-Beta superfamily gene polymorphisms - specifically bone morphogenic protein receptor II, and CORIN, the serine protease which, cleaves the natriuretic peptide precursors secreted by the heart, proANP and proBNP, to the physiologically active ANP and BNP). Finally, our study using the SELDI-TOF-MS system and 2D differential gel electrophoresis (DIGE), will examine differential patterns of plasma protein expression, in particular the apolipoproteins and arginase I and II enzymes, as potential biomarkers or therapeutic targets in sickle cell patients with pulmonary hypertension. Our proposal uniquely integrates international clinical, epidemiologic and molecular studies to determine the burden of SCD related PAH, decipher the mechanism of interactions of PAH and infectious diseases and identify genetic and protein markers and potential therapeutic targets for PAH. Our collaboration will provide an opportunity for the rapid transfer of appropriate technology and knowledge relevant to the provision of the highest quality care to sickle cell patients in Nigeria and the world.

ELIGIBILITY:
* INCLUSION CRITERIA:

All volunteer subjects 5 years of age and above and able to provide informed, written consent for participation in this study. Children will be included in this study provided that a legally authorized representative provides fully informed consent. Assent of children will also be required.

Inclusion Criteria for Volunteers with Sickle Cell:

* Nigerian male and females over 5 years of age
* Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, or SBeta thalassemia or other genotype is required)

Inclusion Criteria for Control Subjects:

* Nigerian males and females over 5 years of age.
* Electrophoretic documentation of hemoglobin A or AS genotype.

EXCLUSION CRITERIA:

Exclusion Criteria for Volunteers with Sickle Cell:

* Hb A-only phenotype and sickle cell trait
* Decisionally impaired subjects.
* Persons not able to understand the investigational nature of the study or give informed consent.

Exclusion Criteria for Control Subjects:

* Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, SBeta thallassemia or other sickling genotype)
* Decisionally impaired subjects.
* Persons not able to understand the investigational nature of the study or give informed consent.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2006-06-15; Study Completion 2017-09-28

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Ahmadu Bello University Teaching Hospital, Kaduna, Nigeria

REFERENCES:
- [Background] Aliyu ZY, Tumblin AR, Kato GJ. Current therapy of sickle cell disease. Haematologica. 2006 Jan;91(1):7-10. No abstract available. PMID 16434364
- [Background] Rother RP, Bell L, Hillmen P, Gladwin MT. The clinical sequelae of intravascular hemolysis and extracellular plasma hemoglobin: a novel mechanism of human disease. JAMA. 2005 Apr 6;293(13):1653-62. doi: 10.1001/jama.293.13.1653. PMID 15811985
- [Background] Morris CR, Kato GJ, Poljakovic M, Wang X, Blackwelder WC, Sachdev V, Hazen SL, Vichinsky EP, Morris SM Jr, Gladwin MT. Dysregulated arginine metabolism, hemolysis-associated pulmonary hypertension, and mortality in sickle cell disease. JAMA. 2005 Jul 6;294(1):81-90. doi: 10.1001/jama.294.1.81. PMID 15998894